CLINICAL TRIAL: NCT00145054
Title: Randomized, Controlled Pilot Study of a Self-Help Depression Skills Program for College-Aged Youth
Brief Title: Study of a Self-Help Depression Skills Program for College-Aged Youth
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R24MH061422 (NIH)
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2006-03-24 (Estimated); Status verified 2005-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

INTERVENTIONS:
Behavioral: MoodHelper Internet program for Depression Self-Help

SUMMARY:
We propose to conduct a pilot trial of an Internet-only depression skills training program for adolescents and young adults. The intervention, MoodHelper.org already exists and has been tested in two pilots. In this third pilot, we plan to use an enriched minority sampling frame to mail 3,000 to 6,000 invitational brochures to KPNW members aged 14 to 24, with a enrollment target of 150. Interested members will go to the study Internet site, and if they choose to participate, complete the online consent and assessment battery (used in the previous pilots). Participants will be randomly assigned by the site's software to one of two conditions: (1) the "Intervention" condition, with complete access to the SADhelper.org web site or (2) the "Usual Care" condition, with access to all Internet sites and KPNW health care, but with no access to the therapeutic portion of the SADhelper site. All participants (those with and without access to the research intervention) will be reminded by e-mail and, if necessary, by telephone to return to the web site and complete follow-up questionnaires four, eight, sixteen, and thirty-two weeks after enrolling in the study.

DETAILED DESCRIPTION:
We propose to conduct a pilot trial of an Internet-only depression skills training program for adolescents and young adults. The intervention, MoodHelper.org already exists and has been tested in two pilots. In this third pilot, we plan to use an enriched minority sampling frame to mail 3,000 to 6,000 invitational brochures to KPNW members aged 14 to 24, with a enrollment target of 150. Interested members will go to the study Internet site, and if they choose to participate, complete the online consent and assessment battery (used in the previous pilots). Participants will be randomly assigned by the site's software to one of two conditions: (1) the "Intervention" condition, with complete access to the SADhelper.org web site or (2) the "Usual Care" condition, with access to all Internet sites and KPNW health care, but with no access to the therapeutic portion of the SADhelper site. All participants (those with and without access to the research intervention) will be reminded by e-mail and, if necessary, by telephone to return to the web site and complete follow-up questionnaires four, eight, sixteen, and thirty-two weeks after enrolling in the study.

ELIGIBILITY:
Inclusion Criteria:

current clinical diagnosis of depression Internet access

Exclusion Criteria:

none

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150

PRIMARY OUTCOMES:
self-reported depression on the CES-D

SECONDARY OUTCOMES:
health care utilization

CONTACTS AND LOCATIONS:
Overall Officials: Greg Clarke, Ph.D., Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

REFERENCES:
- [Derived] Clarke G, Kelleher C, Hornbrook M, Debar L, Dickerson J, Gullion C. Randomized effectiveness trial of an Internet, pure self-help, cognitive behavioral intervention for depressive symptoms in young adults. Cogn Behav Ther. 2009;38(4):222-34. doi: 10.1080/16506070802675353. PMID 19440896